CLINICAL TRIAL: NCT03361436
Title: A Phase 1B Trial of Preoperative Eribulin and Radiation for Retroperitoneal Liposarcoma
Brief Title: Eribulin and Radiation Therapy in Treating Patients With Retroperitoneal Liposarcoma That Can Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Eisai Inc. (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Lara Davis, MD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00017190; NCI-2017-02120 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00017190 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Liposarcoma; Malignant Abdominal Neoplasm; Malignant Retroperitoneal Neoplasm; Malignant Scrotal Neoplasm; Malignant Solid Neoplasm; Malignant Spermatic Cord Neoplasm
MeSH Terms: conditions — Liposarcoma | interventions — eribulin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (eribulin mesylate, IMRT, surgery) (Experimental): Patients receive eribulin mesylate IV over 2-5 minutes on days 1 and 8 and undergo intensity-modulated radiation therapy QD 5 days a week beginning on day 8 of cycle 1. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients may undergo surgery within 3-10 weeks after radiation therapy.
  Interventions: Drug: Eribulin Mesylate; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Eribulin Mesylate — Given IV
  Other Names: B1939 Mesylate; E7389; ER-086526; Halaven; Halichondrin B Analog
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase Ib trials studies the side effects and best dose of eribulin mesylate when given together with radiation therapy in treating patients with retroperitoneal liposarcoma that can be removed by surgery. Drugs used in chemotherapy, such as eribulin mesylate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving chemotherapy with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase 2 dose (RP2D) of radiation and eribulin mesylate (eribulin) when used in combination for the preoperative treatment of retroperitoneal liposarcoma.

SECONDARY OBJECTIVES:

I. To assess the feasibility of a preoperative chemoradiation protocol for retroperitoneal liposarcoma.

II. To assess the surgical outcomes of retroperitoneal liposarcoma resections after preoperative chemoradiation.

III. To assess preliminary anti-tumor activity of eribulin in combination with radiation in subjects with retroperitoneal liposarcoma.

OUTLINE: This is a dose-escalation study of eribulin mesylate.

Patients receive eribulin mesylate intravenously (IV) over 2-5 minutes on days 1 and 8 and undergo intensity-modulated radiation therapy once daily (QD) 5 days a week beginning on day 8 of cycle 1. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients may undergo surgery within 3-10 weeks after radiation therapy.

After completion of study treatment, patients will be followed up at 2 weeks, 9 weeks, and then every 6 months for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of liposarcoma; all subtypes are eligible
* Sufficient archival tissue available for correlative studies; submission of formalin-fixed paraffin-embedded (FFPE) tumor tissue from a previous biopsy or resection is required, and the most recent specimen is preferred; if a FFPE block cannot be provided, then 10 unstained, positively-charged slides of 4-5 um thickness must be submitted; if insufficient archival tissue is available, a repeat biopsy will be necessary
* Primary or recurrent retroperitoneal, scrotal/spermatic cord or abdominal tumor
* For subjects between the ages of 12-18 years only, body surface area (BSA) must be >= 1.5 m^2
* All sites of disease must be resectable or borderline resectable as assessed by a surgical oncologist with experience in retroperitoneal sarcoma resection after discussion in our institutional multidisciplinary sarcoma tumor board conference
* All sites of disease must be targetable with intensity-modulated radiation therapy (IMRT) with acceptable morbidity and without exceeding normal tissue dose constraints as assessed by a radiation oncologist
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Subjects of childbearing potential must have a negative urine beta-human chorionic gonadotropin (beta-hCG) pregnancy test at time of screening
* Fridericia's correction formula (QTcF) interval on standard 12-lead electrocardiography (ECG) parameters at screening (defined as the mean of the triplicate ECGs) of < 450 msec for males and < 470 msec for females
* Ejection fraction of >= 50%
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Individuals of childbearing potential must be willing to use adequate contraception throughout the study and for 3 weeks after study drug discontinuation
* Absolute neutrophil count (ANC) >= 1 K/cu mm
* Platelets (no transfusion within prior 7 days) >= 100 K/cu mm
* Hemoglobin (no transfusion within prior 7 days) >= 9.0 g/dL
* Total bilirubin < institutional upper limit of normal (ULN), except for subjects with documented Gilbert's syndrome, for which =< 3.0 x ULN or direct bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Estimated creatinine clearance > 50 mL/min by Cockcroft-Gault equation
* Ability to understand and the willingness to sign a written informed consent document; subject has signed the informed consent (ICF) prior to any screening procedures being performed and is able to comply with protocol requirements

Exclusion Criteria:

* Presence of distant metastases; intra-abdominal (regional) spread is allowable if meets inclusion criterial indeterminate or small volume pulmonary nodules may be eligible, if the treating physicians recommend curative-intent resection of the primary tumor despite the presence of possible lung metastases
* Prior radiation or systemic therapy for the diagnosis of liposarcoma
* Prior eribulin
* Grade >= 2 peripheral neuropathy
* Contraindication to magnetic resonance imaging (MRI), including presence of a pacemaker or aneurysm clip, severe claustrophobia, a known reaction to gadolinium contrast, or body weight exceeding 300 pounds (lbs)
* Concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of malignancies that have completed therapy and are considered by their physician to be at less than 30% risk of relapse; prior systemic therapy is allowed with the exception of prior eribulin; prior radiation therapy is allowed with the exception of any abdominal, pelvic or retroperitoneal radiation > 10 Gy
* History of uncontrolled arrhythmia, congenital long QT syndrome or torsades de pointes (TdP)
* Use of more than one medication with a known risk of TdP
* Major operation within 14 days prior to starting study drug or not recovered from surgical complications; neither tumor biopsy nor central line insertion are considered a major operation
* Active infection; any systemic antimicrobial therapy must be completed >= 5 days prior to initiation of protocol therapy
* Pregnant or nursing (lactating) individuals; NOTE: Pregnant individuals are excluded from this study because eribulin is an investigational agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the individual with eribulin breastfeeding should be discontinued; these potential risks may also apply to doxorubicin
* Unable or unwilling to stop the use of herbal supplements; the use of marijuana or its derivatives is allowed; the use of supplements may be allowed after review by a study pharmacist to confirm no significant risk of interaction with eribulin or radiation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2033-04-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities according to Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03 | Up to 42 days
  All adverse events will be tabulated and summarized by major organ category, grade, anticipation, and drug attribution. Serious adverse events (SAE) specific incidence and exact 95% confidence interval will be provided where appropriate.

SECONDARY OUTCOMES:
Rate of enrollment | Up to 18 months
Rate of early surgical resection | 3 weeks after radiation therapy
  The proportion of subjects, along with exact two-sided 95% confidence intervals, undergoing surgical resection before the completion of all planned chemotherapy and radiation will be reported for the study.
Rate of surgical resection | After 10 weeks of radiation, until study completion (up to 4 years)
  The proportion of subjects, along with exact two-sided 95% confidence intervals, undergoing surgical resection later than planned for any reason will be reported for the study.
Change in subject-reported quality of life assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline up to 9 weeks after surgery
  Will apply a mixed effects model to analyze changes in PROMIS symptom measurements at four time points: baseline, C2D8, prior to surgery and 9 weeks postoperative (post-op).
Rate of R0 resection defined as the proportion of surgical specimens with microscopically negative margins | Up to 10 years
  The rate of R0 resection, along with exact two-sided 95% confidence intervals, will be reported for the study.
Rate of serious post-operative complications | Up to 9 weeks following surgery
  This rate, along with exact two-sided 95% confidence intervals, will be reported for the study.
Pathologic response defined as the percentage of tumor with treatment change, including necrosis, fat maturation and hyalinization | Up to 10 years
  Descriptive statistics including mean, median, standard deviation, and 95% confidence interval of pathologic response will be reported for the study.
Objective response rate (ORR) defined as the proportion of subjects who achieved a complete response (disappearance of all target tumors) or a partial response (>= 30% decrease in the sum of the longest diameters of target tumors) | Up to 10 years
  Based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The ORR, along with exact two-sided 95% confidence intervals, will be reported for the study.
Recurrence-free survival rate | Up to 10 years
  Median recurrence-free survival with 95% confidence interval (CI) and survival rates at 2, 5 and 10 years will be estimated using the Kaplan-Meier method for both local and distant recurrence.
Overall survival rate | Up to 10 years
  Median overall survival with 95% CI and survival rates at 2, 5 and 10 years will be estimated using Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Lara E Davis, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vatner R, James CD, Sathiaseelan V, Bondra KM, Kalapurakal JA, Houghton PJ. Radiation therapy and molecular-targeted agents in preclinical testing for immunotherapy, brain tumors, and sarcomas: Opportunities and challenges. Pediatr Blood Cancer. 2021 May;68 Suppl 2:e28439. doi: 10.1002/pbc.28439. Epub 2020 Aug 22. PMID 32827353